CLINICAL TRIAL: NCT06355115
Title: Comparison Effect Between a Single Dose Prophylaxis Antibiotics Given One Day and Three Days Towards Healing and Risk of Infection in Permanent Pacemaker (PPM) Installation: a Preliminary Study
Brief Title: Prophylactic Antibiotics Duration Towards Healing and Risk of Infection in Permanent Pacemaker (PPM) Installation
Acronym: PACE-PRO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Brawijaya (Other)
Collaborators: Saiful Anwar Hospital (Other)
Responsible Party: Principal Investigator, Icmi Dian Rochmawati, Clinical Cardiologist, University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 400/218/K.3/302/2023
Record Dates: First submitted 2023-12-19; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pacemaker Complication
Keywords: permanent pacemakers; infections; prophylactic antibiotics
MeSH Terms: conditions — Infections | interventions — Cefazolin; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Three days dose prophylaxis (Active Comparator): Intravenous (iv) injection of Cefazolin 1 gram 1-hour pre-procedure followed by iv injection of Cefazolin 1 gram every 12 hours for 3 days post-procedure (6 doses)
  Interventions: Drug: Cefazolin 1000 MG Injection
- Single dose prophylaxis (Experimental): Intravenous injection of Cefazolin 1 gram 1-hour pre-procedure
  Interventions: Drug: Cefazolin 1000 MG Injection

INTERVENTIONS:
Drug: Cefazolin 1000 MG Injection — Cefazolin 1000 mg given intravenously

SUMMARY:
The insertion of a permanent pacemaker (PPM) is frequently a life-saving procedure. However, the implantation process could sometimes lead to a rare but serious infection. Therefore, administering prophylactic antibiotics to prevent infections before they occur, is a useful strategy to lower the risk of such infections.

Nonetheless, the optimal duration of prophylactic antibiotics for PPM remains uncertain. Individual study results are ambiguous and debatable due to the fact that each center has its own policy governing the regimen for prophylactic antibiotic use. Accordingly, the goal of this clinical trial is to assess and compare the effectiveness of two types of widely used prophylactic antibiotic durations in relation to the risk of infections following PPM implantations.

The main questions it aims to answer are:

1. What is the efficacy of different durations of prophylactic antibiotics (single dosage vs 3-day dosage) in preventing infective complications following PPM implantations?
2. What factors may influence the optimum use of prophylactic antibiotics for individual patients undergoing PPM implantation to minimize the risk of infective complications?

Researchers will compare a single dosage vs a 3-day dosage of prophylactic antibiotics following the PPM implantation procedure to see the risk of device-related infections.

Participants will:

* Be given a single-dose or 3-days dose of antibiotic regarding the PPM installations.
* Visit the clinic for follow-ups and tests.

DETAILED DESCRIPTION:
The insertion of a permanent pacemaker (PPM) is a critical intervention often performed to manage various cardiac rhythm disorders, thereby enhancing patient survival and quality of life. However, the procedure carries a risk of introducing infections, which, although infrequent, can lead to severe complications. Prophylactic administration of antibiotics has been recognized as an effective measure to mitigate this risk by preventing the onset of infections prior to their occurrence.

Despite the widespread acceptance of this practice, the optimal duration of antibiotic prophylaxis for PPM implantation remains a subject of debate. Variability in clinical protocols across different healthcare centers further complicates the establishment of a standardized approach. This clinical trial is designed to address this gap by evaluating and comparing the efficacy of two commonly employed prophylactic antibiotic regimens - a single dose versus a three-day course - in reducing the incidence of infectious complications following PPM implantations.

The study aims to address the following research questions:

1. What is the comparative effectiveness of a single dose versus a three-day course of prophylactic antibiotics in preventing infectious complications after PPM implantation?
2. What patient-specific or procedural factors might influence the optimal choice and duration of prophylactic antibiotic therapy in the context of PPM implantation?

To achieve these objectives, the trial will enroll patients scheduled for PPM implantation and randomly assign them to receive either a single dose or a three-day course of antibiotics. The choice of antibiotic will be based on our institutional guidelines, i.e. 1 gram of intravenous Cefazolin (first-generation cephalosporins), and by considering the patient's allergy history. The primary outcome will be the occurrence of device-related infections within a specified follow-up period, assessed through clinical examinations, laboratory tests, and imaging studies.

Participants will be required to attend follow-up visits at designated intervals post-implantation for assessment of any signs of infection, wound healing, and device function. Adherence to the antibiotic regimen and any adverse reactions will also be monitored.

By systematically comparing the outcomes of the two antibiotic regimens, this study aims to provide evidence-based guidance for the optimization of prophylactic antibiotic use in PPM implantations, thereby enhancing patient safety and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

Case inclusion criteria

1. Adult patients, aged 18 to 100 years old, with indications for PPM (single or double chamber) installation.
2. The patient is scheduled to undergo PPM installation for the first time
3. The patient is willing to undergo routine follow-ups and visits
4. Patients who are medically stable and do not have any acute illnesses that could interfere with the study outcomes.

Exclusion Criteria:

1. Patients with fever before the Procedure
2. Skin disease
3. Patients on anticoagulants or receiving bridging heparin
4. Patients who used antibiotics 30 days before the PPM installation was carried out
5. Patients with end stage renal failure
6. Patients with uncontrolled Diabetes Mellitus
7. Patients with a history of infective endocarditis
8. Patients with a history of moderate to severe valvular heart disease
9. Patients with congenital heart disease
10. Patients with non-cardiac comorbid diseases whose life expectancy is < 1 year
11. Illness or physical disorder that causes the patient to be unable or limited to carry out physical activities
12. Patients with a history of autoimmune disease, and confirmed autoimmune disease
13. Patients on long-term steroid use
14. The patient refused follow-up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with early pocket infection (EPI) | 0-30 days
  EPI refers to a post-operative complication characterized by wound infection or infection of the device pouch within the initial weeks or month following surgical procedure. Manifestations of early pocket infections include local signs of inflammation such as erythema, edema, warmth, and tenderness at the implantation site, occasionally accompanied by purulent discharge or systemic symptoms such as fever.
Number of participants with late pocket infection (LPI) | 1-3 months
  LPI refers to a post-operative complication characterized by wound infection or infection of the device pouch within the following months following surgical procedure. Manifestations of late pocket infections are similar to those of EPI, which include local signs of inflammation such as erythema, edema, warmth, and tenderness at the implantation site, occasionally accompanied by purulent discharge or systemic symptoms such as fever.
Number of participants with infective endocarditis (IE) | 1 year
  IE following the implantation of PPM is characterized by bacteremia due to device infection, lead vegetation, right infective endocarditis. Diagnosis is established through history taking and physical examination and the visualization of vegetations by Transthoracic Echocardiography (TTE).
Number of participants who underwent pacemaker revision | 1 year
  Pacemaker revision or reimplantation due to infective complications.

SECONDARY OUTCOMES:
Level of C-reactive protein (mg/dl) | 3 days
  C-reactive protein (CRP) levels will be measured from venous blood samples obtained from patients on the third day following the PPM implantation procedure.
Level of procalcitonin (mcg/dl) | 3 days
  Procalcitonin (PCT) levels will be measured from venous blood samples obtained from patients on the third day following the PPM implantation procedure.
Erythrocyte sedimentation rate (ESR) (mm/hour) | 3 days
  Erythrocyte sedimentation rate (ESR) levels will be measured from venous blood samples obtained from patients on the third day following the PPM implantation procedure.
Neutrophil-to-leukocyte ratio (NLR) | 3 days
  Neutrophil-to-leukocyte ratio (NLR) levels will be measured from venous blood samples obtained from patients on the third day following the PPM implantation procedure.
Neutrophil count (cells/mm3) | 3 days
  Neutrophil count levels will be measured from venous blood samples obtained from patients as part of complete blood count testing, on the third day following the PPM implantation procedure.
Leukocyte count (cells/mm3) | 3 days
  Leukocyte (white blood cells) count levels will be measured from venous blood samples obtained from patients as part of complete blood count testing, on the third day following the PPM implantation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Icmi D Rochmawati, M.D., Principal Investigator — University of Brawijaya
Locations (1):
- RSUD Dr. Saiful Anwar, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Access to the collected data will be restricted solely to authorized members of the research team.